CLINICAL TRIAL: NCT03936491
Title: The Neuroprotective Effects of Methylphenidate and Atomoxetine in Children With Attention Deficit Hyperactivity Disorder: A Lipidomic Study
Brief Title: The Neuroprotective Effects of Methylphenidate and Atomoxetine in Children With ADHD: A Lipidomic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812200MINA
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: biomarker; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate (Experimental): The subjects will receive methylphenidate according to their clinical symptoms
  Interventions: Drug: Methylphenidate
- Atomoxetine (Active Comparator): The subjects will receive atomoxetine according to their clinical symptoms
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate is a central nervous system stimulant used for the therapy of attention deficit disorder and narcolepsy.
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Atomoxetine — Atomoxetine is a medication used to treat attention deficit hyperactivity disorder (ADHD).[6] Use is only recommended in those who are at least six years old.[6] It is taken by mouth.[6]
  Other Names: Strattera
  Arms: Atomoxetine

SUMMARY:
1. To identify the difference in the lipidomic profiles between ADHD and controls;
2. To examine the effects of methylphenidate and atomoxetine on the lipidomic profiles in ADHD, and the relationship between medication-related changes in the lipidomic profiles and medication-related improvements in the behavioral symptoms and neuropsychological functions;
3. To map medication-related lipidomic biomolecules to their respective metabolic pathways to identify the underlying mechanisms of neuroprotective effects of methylphenidate and atomoxetine.

DETAILED DESCRIPTION:
Background: Although the efficacy of methylphenidate and atomoxetine in ADHD is well documented in clinical trials, more studies are needed to clarify the neuroprotective effects of these two medications. Lipids exert important neuroprotective effects for optimal brain development and functioning. Previous studies have demonstrated the significant connection between lipid dysregulation and the occurrence of ADHD. In addition, lipid dysregulation is closely related to the abnormal neural activity in individuals with ADHD. In this 3-year prospective project, we will perform a lipidomic analysis of blood before and after treatment with methylphenidate or atomoxetine, in order to identify the biological connections between the neuroprotective effects of medications and pathways of lipid metabolism in children with ADHD.

Subjects and Methods: 70 drug-naïve patients with ADHD, aged 6-18, and 35 matched typically developing controls will be recruited in this project. We will randomly assign the 70 ADHD patients to two groups, 35 in the methylphenidate group and 35 in the atomoxetine group. Within the 12-week treatment period, we will use ADHDRS-IV, SNAP-IV, CBCL, YSR, CGI-ADHD-S, CGI-ADHD-I, SAICA, and Family APGAR-C to assess the improvement in the behavioral symptoms, and CPT and CANTAB to assess the improvement in the neuropsychological functioning. The blood sample will be collected, and we will use mass spectrometry to assess the medication-related change in lipidomic profiles.

Anticipated Results: Using a prospective design, we anticipate that this study will delineate the effects of methylphenidate and atomoxetine on the lipidomic profiles in patients with ADHD. Furthermore, we will conduct pathway analysis to obtain crucial insight to the lipidomic regulation in neurophysiology of children with ADHD. We expect that the findings will increase our understanding of the neuroprotective effects of methylphenidate and atomoxetine in patients with ADHD, and identify the psychopharmacological mechanism of medication effects in ADHD via the pathways of lipid metabolism and regulation.

ELIGIBILITY:
Subjects will be recruited in the present project if they meet the following inclusion criteria:

1. Children or adolescents, between 6 and 18 years of age, must have ADHD based on the diagnostic criteria of the Diagnostic and Statistical Manual of Mental disorders, 5th edition.
2. Their scores of Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) is greater than 4 at baseline.
3. They have to be medication-naïve. They never receive any medication for the treatment of ADHD.
4. They and their parents must understand sufficiently to communicate properly with the investigators.
5. They must have a Full-Scale Intelligence Quotient (FIQ) score greater than 80.
6. They must keep regular clinic visits and all required tests, including collection of blood sample and neuropsychological testing.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale-IV-Parent version: Investigator-Administered and Scored (ADHDRS-IV) | 12 weeks
  The first efficacy measure is the ADHDRS-IV, which is a scale composed of 18 items. The investigator will conduct a semi-structured interview with the parent to evaluate the severity of ADHD symptoms in the past week. ADHDRS-IV is a valid and reliable tool to assess the severity of ADHD symptoms, which has been widely used in pharmacological studies of ADHD in Taiwanese populations. ADHDRS-IV will be administered from visit 1 through visit 5 (baseline-week 12).

SECONDARY OUTCOMES:
Swanson, Nolan, and Pelham IV scale (SNAP-IV), Parent Form and Teacher Form | 12 weeks
  The SNAP-IV is composed of the ADHD symptoms for the inattention (Items 1 to 9), the hyperactivity/impulsivity (Items 10 to 18), and the oppositional symptoms (Items 19 to 26). SNAP-IV has been proved to be a valid and reliable tool to evaluate the severity of ADHD symptoms. The Chinese SNAP-IV has been used widely in the pharmacological studies on ADHD in Taiwanese populations. SNAP-IV will be administered from visit 1 through visit 5 (baseline-week 12).

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang Shang, MDPHD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan